CLINICAL TRIAL: NCT06901271
Title: The Effect of EMLA Cream, Cold Spray, and Buzzy on Venipuncture Pain and Fear in Children: a Randomized Controlled Trial
Brief Title: Pharmacological and Nonpharmacological Methods for Children in Venipuncture Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aynur Aytekin Ozdemir (Other)
Responsible Party: Sponsor-Investigator, Aynur Aytekin Ozdemir, Professor, Istanbul Medeniyet University
Organization: Istanbul Medeniyet University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018-3/19
Record Dates: First submitted 2025-03-24; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Procedural Pain Relief; Fear Pain
Keywords: Procedural pain; venipuncture; children
MeSH Terms: conditions — Pain, Procedural | interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Intervention Model Description: This study was conducted as a randomized controlled trial in parallel groups. The variables used for blocking were age (7-9 and 10-12 years), sex (female and male), and fear of the procedure (yes and no). The blocks were repeated six times in each group (2 × 2 × 2 × 6 ), resulting in 48 participants per group.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control Group (No Intervention): The control group received the routine venipuncture procedure.
- Intervention 1 Group (Experimental): In this group, EMLA cream was applied to the procedure area (antecubital region) 60 minutes before the venipuncture procedure. Then, the venipuncture procedure was performed.
  Interventions: Drug: EMLA Cream
- Intervention 2 Group (Experimental): In this group, cold spray was applied to the procedure area for 5 seconds just before the venipuncture procedure. Then, the venipuncture procedure was performed.
  Interventions: Drug: Cold spray
- Intervention 3 Group (Experimental): In this group, Buzzy was placed in the procedure area. Buzzy was operated for 60 seconds. Then, the venipuncture procedure was performed. It also operated during this procedure.
  Interventions: Device: Buzzy

INTERVENTIONS:
Drug: EMLA Cream — EMLA cream (2.5 grams) was applied to the treatment area 60 minutes before the procedure and covered with a transparent and impermeable dressing.
  Arms: Intervention 1 Group
Device: Buzzy — The buzzy device was placed on the procedure area 60 seconds before the procedure and turned on. The cold and vibration application continued during the procedure.
  Arms: Intervention 3 Group
Drug: Cold spray — Cold spray was applied to the procedure area for 5 seconds from a distance of 15 cm immediately before the procedure.
  Arms: Intervention 2 Group

SUMMARY:
This study aimed to examine the effect of EMLA cream, cold spray, and Buzzy applied during venipuncture on the pain and fear levels of children aged 7-12 years.

DETAILED DESCRIPTION:
The International Guide to Pediatric Anesthesia (Good Practice in Postoperative and Procedural Pain) recommends pharmacological and nonpharmacological methods to effectively manage and prevent acute procedural pain in children. Nonpharmacological methods alone or in combination with pharmacological methods help reduce pain, and therefore, have become popular especially in recent years. For pain management, nonpharmacological methods are easy to use, and cost- and time-effective methods with no side effects. Studies have evaluated a large number of pharmacological and nonpharmacological interventions for procedural pain management in children. However, most of those interventions are not used by healthcare professionals because they are expensive, time-consuming or hard to use. Therefore, easy-to-use, practical, non-invasive, cost-effective, and reusable pharmacological and nonpharmacological methods can be used especially in acute settings. EMLA cream, cold spray, and Buzzy examined in this study may serve as alternative effective pharmacological and non-pharmacological methods to reduce venipuncture pain and fear.

ELIGIBILITY:
Inclusion Criteria:

* being between the ages of 7 to 12 years,
* literate,
* requiring blood tests

Exclusion Criteria:

* having chronic diseases,
* hospital stay for treatment,
* visual, audio, or speech impairments,
* a history of allergies,
* mental disorders,
* history of sedative, analgesic, or narcotic use within 24 h before admission,
* inflammatory disease during admission.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Procedural pain score- Visual Analog Scale (VAS) | Through painful procedure completion, an average of 5 minutes
  The VAS is used to measure and monitor pain intensity. VAS is a 10 cm or 100 mm long horizontal or vertical line with anchor statements "no pain or pain at its least" at the left-most end and "unbearable pain or worst pain imaginable" at the right-most end. The participant is asked to mark a point on the line that best represents their pain level. The VAS score is determined by measuring the distance of the mark from the left end of the line. VAS is an easy-to-understand and easy-to-measure scale for children aged 7 and over
Procedural pain score- Wong-Baker FACES Pain Rating Scale | Through painful procedure completion, an average of 5 minutes
  The scale is used to diagnose pain in children aged 3-18 years. It consists of six facial expressions, each one representing an increasing degree of pain scored on a scale 0 to 5 from left to right. The first face is a happy face representing "no pain=0" while the last face is a crying face representing "the worst pain imaginable=5". Higher scores indicate low pain tolerance. Participants are asked to choose the facial expression that best represents their pain.

SECONDARY OUTCOMES:
Procedural fear score- Children's Fear Scale (CFS) | Through painful procedure completion, an average of 5 minutes
  The CFS was developed to measure fear and anxiety in children. It consists of five facial expressions that represent a range from neutral to extreme fear. It is scored between 0 and 4. Both researchers and family members can use the CFS to measure fear and anxiety in children before and during procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Aytekin Ozdemir, Professor, Principal Investigator — İstanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be shared upon request from the principal investigator, subject to the appropriateness of the request, while ensuring adherence to the rules of confidentiality regarding individual data.
Supporting Information: Study Protocol
Time Frame: July through December of 2026
Access Criteria: Individual participant data may be shared upon request from the principal investigator, subject to the appropriateness of the request, while ensuring adherence to the rules of confidentiality regarding individual data.

REFERENCES:
- [Background] Dalvandi A, Ranjbar H, Hatamizadeh M, Rahgoi A, Bernstein C. Comparing the effectiveness of vapocoolant spray and lidocaine/procaine cream in reducing pain of intravenous cannulation: A randomized clinical trial. Am J Emerg Med. 2017 Aug;35(8):1064-1068. doi: 10.1016/j.ajem.2017.02.039. Epub 2017 Feb 27. PMID 28285862
- [Background] Celik EG, Sonmez Duzkaya D. The Impact of Cold Spray and Ice Application During Intravenous Access on Pain and Fear in Children Aged 7-15 Years in the Pediatric Emergency Unit: A Randomized Controlled Trial. J Emerg Nurs. 2024 Mar;50(2):264-272. doi: 10.1016/j.jen.2023.11.012. Epub 2023 Dec 24. PMID 38142386
- [Background] Erdogan B, Aytekin Ozdemir A. The Effect of Three Different Methods on Venipuncture Pain and Anxiety in Children: Distraction Cards, Virtual Reality, and Buzzy(R) (Randomized Controlled Trial). J Pediatr Nurs. 2021 May-Jun;58:e54-e62. doi: 10.1016/j.pedn.2021.01.001. Epub 2021 Jan 21. PMID 33485746